CLINICAL TRIAL: NCT00919308
Title: Simulation Training for Ultrasound Guided Central Venous Catheter Insertion
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Leigh V. Evans MD, Yale University School of Medicine
Other Study IDs: 0605001388; 5U18HS016725-02 (AHRQ)
Record Dates: First submitted 2009-06-09; First posted 2009-06-12 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2009-06

CONDITIONS: Procedural Skill Competency
Keywords: Simulation; Invasive procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control, traditional bedside training: Postgraduate year 1 and 2 residents who are trained in central venous catheter insertion according to the traditional, bedside apprenticeship model.
- Simulation training: Postgraduate year 1 and 2 residents who complete a hands-on ultrasound guided simulation training protocol on a partial task training simulator until competence is achieved as measured by: the ability to cannulate a simulated vein under ultrasound guidance on first pass in five consecutive attempts and correct insertion of a central venous cannulator on a partial task training simulator with no technical errors.
  Interventions: Other: Competency based simulation training

INTERVENTIONS:
Other: Competency based simulation training — Completion of a hands-on ultrasound guided simulation training protocol on a partial task training simulator until competence is achieved as measured by the ability to cannulate a simulated vein under ultrasound guidance on first pass in five consecutive attempts and correct insertion of a central venous catheter on a partial task training simulator with no technical errors.
  Groups: Simulation training

SUMMARY:
Hypothesis #1: Residents who complete a structured, ultrasound guided simulation training protocol will have superior skills at central venous catheter (CVC) insertion on actual patients as compared to residents who are trained in CVC insertion according to the traditional, bedside apprenticeship model as measured by a reduced failure rate at CVC insertion.

Hypothesis #2: Residents who complete a structured, ultrasound guided simulation training protocol will have superior skills at CVC insertion on actual patients as compared to residents who are trained in CVC insertion according to the traditional, bedside apprenticeship model as measured by:

1. a reduced number of attempts at venous cannulation,
2. a decreased rate of technical errors and a decreased complication rate based on an independent rater's evaluation using a procedure checklist, and
3. a decreased time to CVC insertion from opening the catheter kit to placement of sterile dressing as timed by an independent rater.

DETAILED DESCRIPTION:
Resident education has traditionally devoted itself to knowledge acquisition rather than defined levels of clinical competence. Currently, inexperienced physicians are trained to perform invasive procedures such as central venous catheter (CVC) insertion according to the bedside, apprenticeship model, gaining expertise on real patients in neither a rigorous nor standardized manner. Simulators may ease trainees' transition to actual patients and avoid adverse events. This project aims to investigate the efficacy of a structured simulation training protocol in ultrasound guided CVC insertion for resident physicians. The specific aims are to compare: (1) the failure rate of CVC insertion, and (2) the number of attempts at venous cannulation, rates of technical errors and complications of CVC insertion, and time to CVC insertion on actual patients between residents who completed a structured, hands-on simulation training protocol (intervention group) and those who are trained according to the traditional, bedside apprenticeship model (control group). We hypothesize that the intervention group will obtain superior skills at CVC insertion on actual patients as compared to the control group as measured by: (1) a reduced failure rate at CVC insertion, (2) a) a reduced number of attempts at venous cannulation b) a decreased rate of technical errors and complications and c) a decreased time to insertion based on an independent rater's evaluation using a procedure checklist.

ELIGIBILITY:
Inclusion Criteria:

Eligibility is determined by the program director of the residency programs.

* The racial, gender, and ethnic characteristics of the proposed subject population reflects the demographics of the interns and residents within the specialties of Emergency Medicine, Internal Medicine, General Surgery, Obstetrics and Gynecology and Anesthesia.
* None of the subjects are minors and all are in sufficient health to participate in their residency programs.

Exclusion Criteria:

* Of eligible subjects, the only exclusion criterion is unwillingness to participate in the project.
* No exclusion criteria shall be based on race, gender, or ethnicity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: PGY-1 or PGY-2 resident status in the Yale-New Haven Hospital Emergency Medicine, Internal Medicine, General Surgery, Obstetric and Gynecology and Anesthesia residency programs.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2006-08; Primary Completion 2008-09 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The failure rate of central venous catheter insertion in the hospital setting on actual patients. | 21 months (January 2007-September 2008)

SECONDARY OUTCOMES:
The number of attempts at venous cannulation, and the rate of technical errors and complication rate of central venous catheter insertion in the hospital setting on actual patients | 21 months (January 2007-September 2008)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Evans LV, Dodge KL, Shah TD, Kaplan LJ, Siegel MD, Moore CL, Hamann CJ, Lin Z, D'Onofrio G. Simulation training in central venous catheter insertion: improved performance in clinical practice. Acad Med. 2010 Sep;85(9):1462-9. doi: 10.1097/ACM.0b013e3181eac9a3. PMID 20736674